CLINICAL TRIAL: NCT05133609
Title: COVID-19 VACCINE SAFETY AND EFFECTIVENESS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Espirito Santo (Other)
Collaborators: Centro de Pesquisas René Rachou (Other Government)
Responsible Party: Principal Investigator, Valéria Valim, Professor, Federal University of Espirito Santo
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: FUES03
Record Dates: First submitted 2021-11-01; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: SARS-CoV-2 Infection
Keywords: vaccines; immunity; safety; rheumatic diseases; covid-19
MeSH Terms: conditions — COVID-19; Rheumatic Diseases | interventions — ChAdOx1 nCoV-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Health professionals who will receive vaccine in the vaccination campaign against SARS-CoV-2.
  Interventions: Biological: ChAdOx1 nCoV-19 vaccine (AZD1222)
- Group 2 (Experimental): Patients with immune-mediated inflammatory diseases who will receive vaccine in the vaccination campaign against SARS-CoV-2.
  Interventions: Biological: ChAdOx1 nCoV-19 vaccine (AZD1222)

INTERVENTIONS:
Biological: ChAdOx1 nCoV-19 vaccine (AZD1222) — ChAdOx1 nCoV-19 vaccine (AZD1222) in a standard 3-dose schedule with an interval of 12 weeks (first-second dose) and 24 weeks (second-third dose).

SUMMARY:
A longitudinal open-label study will include health professionals and patients with immune-mediated inflammatory diseases (IMID) who will receive the ChAdOx1 nCoV-19 vaccine (AZD1222), in a standard 3-dose schedule with an interval of 12 weeks (first-second dose) and 24 weeks (second-thrid dose), in the vaccination campaign against SARS-CoV-2 to assess the safety, efficacy and duration of the short- and long-term humoral and cellular immune response after vaccination for COVID-19 and compare the vaccine response between individuals who have or have not had previous SARS-Cov 2 infection.

DETAILED DESCRIPTION:
A longitudinal open-label study that will include individuals who will receive the ChAdOx1 nCoV-19 vaccine (AZD1222), in a standard 3-dose schedule with an interval of 12 weeks (first-second dose) and 24 weeks (second-thrid dose), in the vaccination campaign against SARS-CoV-2 to assess the safety, efficacy and duration of the short- and long-term humoral and cellular immune response after vaccination for COVID- 19 and compare the vaccine response between individuals who have or have not had previous SARS-Cov 2 infection. Health professionals (HS) and patients with immune-mediated inflammatory diseases (IMID) who participate in vaccination campaigns at the Cassiano Antônio Mores da University Hospital will be included. Federal University of Espírito Santo (HUCAM-UFES). It is intended to include 200 health workers and 350 patients with IMID, totaling 550 participants. Participants who have had previous SARS-CoV-2 infection confirmed by RT-PCR or positive PRNT at baseline will be considered a group exposed to COVID-19 (CovPrev) and the group without previous infection will be considered a control group (Naive). The IMID group will include patients with Rheumatoid Arthritis (RA), Systemic Lupus Erythematosus (SLE), Spondyloarthritis (SA), Sjögren's Syndrome (SS), Psoriasis (Pso), Inflammatory Bowel Disease (IBD) and Vasculitis (VASC) who complete validated international classification criteria for each disease. The criteria for vaccination in the IMID group will be in accordance with the National Immunization Program of the Ministry of Health (PNI/MS). Adverse events will be recorded during the first, second and fourth week, and through weekly telephone contacts until D40. The evaluations and collection of biological samples will be carried out in 5 moments (D0, D14 and D28 after the first dose; D28 after the second dose; and D28 after thrid dose) to evaluate the efficacy and in 3 moments (D180, D360 and D540), to evaluate the duration of immunity. Neutralization tests by plaque reduction (PRNT) will be performed to detect neutralizing antibodies against COVID-19, determination of the profile of specific IgM, IgA and IgG, dosage of systemic soluble factors (chemokines, cytokines and growth factors), characterization of phenotypes of immunoregulation, immunosenescence, cell activation and exhaustion and antigen-specific stimulation of peripheral blood mononuclear cells in vitro. The study hypothesis is that vaccine-induced production of neutralizing antibodies is more effective in individuals with previous natural SARS-Cov2 infection and less in immunosuppressed individuals.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older

Exclusion Criteria:

* Pregnant women;
* History of severe adverse reaction to any previously administered vaccine;
* Having received another vaccine in the last 30 days.

  * The criteria for vaccination in the immune-mediated inflammatory diseases (IMID) group will be in accordance with the Ministry of Health's National Immunization Program (PNI/MS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Viral Neutralization Assay | 7 months
  Neutralizing antibody titers will be expressed by the ability of antibodies to neutralize up to 50% the number of plaques (PRNT50). Title > 1:50 will be considered positive.
Viral Neutralization Assay | 24 months
  Neutralizing antibody titers will be expressed by the ability of antibodies to neutralize up to 50% the number of plaques (PRNT50). Title > 1:50 will be considered positive.

SECONDARY OUTCOMES:
IgM (Immunoglobulin M) | 7 months
  Determination of specific IgM profile. Results will be expressed in fluorescence intensity or pg/ml.
IgM (Immunoglobulin M) | 24 months
  Determination of specific IgM profile. Results will be expressed in fluorescence intensity or pg/ml.
IgG (Immunoglobulin G) | 7 months
  Determination of specific IgG profile. Results will be expressed in fluorescence intensity or pg/ml.
IgG (Immunoglobulin G) | 24 months
  Determination of specific IgG profile. Results will be expressed in fluorescence intensity or pg/ml.
IgA (Immunoglobulin G) | 7 months
  Determination of specific IgA profile. Results will be expressed in fluorescence intensity or pg/ml.
IgA (Immunoglobulin G) | 24 months
  Determination of specific IgA profile. Results will be expressed in fluorescence intensity or pg/ml.
systemic soluble factors | 7 months
  Dosage of soluble systemic factors (chemokines, cytokines and growth factors). Results will be expressed in pg/ml.
systemic soluble factors | 24 months
  Dosage of soluble systemic factors (chemokines, cytokines and growth factors). Results will be expressed in pg/ml.
Antigen-specific stimulation of peripheral blood mononuclear cells | 1 month
  Antigen-specific stimulation of peripheral blood mononuclear cells in vitro. The results will be expressed in percentage positive frequency for a specific cell phenotype.
Antigen-specific stimulation of peripheral blood mononuclear cells | 6 months
  Antigen-specific stimulation of peripheral blood mononuclear cells in vitro. The results will be expressed in percentage positive frequency for a specific cell phenotype.
Antigen-specific stimulation of peripheral blood mononuclear cells | 12 months
  Antigen-specific stimulation of peripheral blood mononuclear cells in vitro. The results will be expressed in percentage positive frequency for a specific cell phenotype.
Antigen-specific stimulation of peripheral blood mononuclear cells | 18 months
  Antigen-specific stimulation of peripheral blood mononuclear cells in vitro. The results will be expressed in percentage positive frequency for a specific cell phenotype.
Lymphocyte investigation | 1 month
  Investigation of memory T and B lymphocytes. The results will be expressed in percentage positive frequency for a specific cell phenotype.
Lymphocyte investigation | 6 months
  Investigation of memory T and B lymphocytes. The results will be expressed in percentage positive frequency for a specific cell phenotype.
Lymphocyte investigation | 12 months
  Investigation of memory T and B lymphocytes. The results will be expressed in percentage positive frequency for a specific cell phenotype.
Lymphocyte investigation | 18 months
  Investigation of memory T and B lymphocytes. The results will be expressed in percentage positive frequency for a specific cell phenotype.
Cytokine investigation | 1 month
  Investigation of intracytoplasmic cytokines. The results will be expressed in percentage positive frequency for a specific cell phenotype.
Cytokine investigation | 6 months
  Investigation of intracytoplasmic cytokines. The results will be expressed in percentage positive frequency for a specific cell phenotype.
Cytokine investigation | 12 months
  Investigation of intracytoplasmic cytokines. The results will be expressed in percentage positive frequency for a specific cell phenotype.
Cytokine investigation | 18 months
  Investigation of intracytoplasmic cytokines. The results will be expressed in percentage positive frequency for a specific cell phenotype.
Adverse events | 1 month
  All adverse events will be followed up to establish severity and causal correlation. There will be surveillance of deaths and will be reported to the ethics committee.
Adverse events | 4 months
  All adverse events will be followed up to establish severity and causal correlation. There will be surveillance of deaths and will be reported to the ethics committee.
Adverse events | 6 months
  All adverse events will be followed up to establish severity and causal correlation. There will be surveillance of deaths and will be reported to the ethics committee.
severe cases of COVID-19 | 24 months
  incidence of severe cases of COVID-19 over 20 months following treatment
deaths | 24 months
  Number of deaths with specific ICD for covid-19
hospital admissions | 24 months
  number of hospital admissions for covid-19
intensive care unit (ICU) admissions | 24 months
  number of intensive care unit (ICU) admissions for the treatment of SARS

CONTACTS AND LOCATIONS:
Overall Officials: Valéria Valim, PhD, Principal Investigator — Federal University of Espirito Santo
Locations (1):
- Federal University of Espirito Santo, Vitória, Espírito Santo, Brazil